CLINICAL TRIAL: NCT04434430
Title: Effectiveness of Preemptive Oral Gabapentin 600 mg on Morphine Requirement After Non Obstetric Lower Abdominal Surgery
Brief Title: Preemptive Oral Gabapentin 600 mg in Reducing Morphine Requirement After Non Obstetric Lower Abdominal Surgery
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Andi Ade Wijaya Ramlan, Principal Investigator, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IndonesiaUAnes 054
Record Dates: First submitted 2020-05-29; First posted 2020-06-16 (Actual); Last update posted 2021-09-13 (Actual); Status verified 2021-09

CONDITIONS: Non-obstetric Lower Abdominal Surgery
Keywords: preemptive analgesia; gabapentin; morphine; lower abdominal surgery
MeSH Terms: interventions — Gabapentin

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gabapentin (Active Comparator): Patient will receive preemptive oral gabapentin 600 mg
  Interventions: Drug: Gabapentin
- Placebo (Placebo Comparator): Patient will receive oral placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Gabapentin — Oral Gabapentin 600 mg
  Arms: Gabapentin
Other: Placebo — Oral NaCl 500 mg
  Arms: Placebo

SUMMARY:
This study aimed to get the information about the effectiveness of preemptive oral gabapentin 600 mg in reducing morphine requirement after non obstetric lower abdominal surgery

DETAILED DESCRIPTION:
Seventy-two subjects were given informed consent before enrolling the study and randomized into two groups; gabapentin and placebo. Two hours before the incision, patients were given preemptive analgesia, either gabapentin or placebo. Non-invasive blood pressure monitor, electrocardiogram (ECG), and pulse oxymetry were set on the subjects in the operating room. General anesthesia induction was done by fentanyl 2 mcg/kg and propofol 2 mg/kg. Endotracheal tube (ETT) intubation was facilitated with atracurium 0.5 mg/kg as muscle relaxant. Maintenance was done by sevoflurane, oxygen, and compressed air. After surgery, patients were extubated until fully conscious. Patients will be transported to recovery room postoperatively. Besides paracetamol as the postoperative analgesia, we also attached patient controlled analgesia (PCA) system to patients' intravenous line using continuous ambulatory delivery device (CADD) contained morphine 1 mg/ml with settings 1 mg per requirement, interval limit within 5 minutes, maximum dose 6 mg/hour intravenously. Cumulative morphine requirement, mean visual analogue scale, and time interval after surgery to the first administration of morphine will be assessed in this study.

ELIGIBILITY:
Inclusion criteria:

* Male or female
* Age: 18-65 years old
* Weigh in range around 20% of the ideal body weight
* Physical status ASA I-II
* Scheduled for elective non-obstetric lower abdominal surgery with general anesthesia
* Duration of surgery less than 4 hours
* Patients who agreed to participate in this study and sign informed consent

Exclusion criteria:

* Patients who have history of allergy or hypersensitivity to gabapentin, paracetamol, morphine, or the other opioids
* Patients who consumed analgesia and NSAID less than 12 hours before surgery
* Patients who experienced physical trauma less than 4 days before surgery
* Patients who have contraindications to gabapentin, morphine, and paracetamol
* Patients who were treated with neuraxial block or peripheral nerve block before and during surgery
* Patients who have history of diabetes, severe live or renal disease
* Patients who were treated with antihypertension, sedatives, hypnotics, antidepressants, and the other drugs that have effects on nervous system
* Patients who have psychiatric disorders
* Patients who consumed gabapentin before perioperative period
* Pregnant or breastfeeding patients

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2019-11-11 (Actual); Primary Completion 2020-02-29 (Actual); Study Completion 2020-02-29 (Actual)

PRIMARY OUTCOMES:
Cumulative morphine requirement within 24 hours after non obstetric lower abdominal surgery | 24 hours after surgery
  Measured by total consumption of morphine on patient controlled analgesia machine
Pain within 24 hours after non obstetric lower abdominal surgerysurgery: visual analogue scale | 24 hours after surgery
  Measured by visual analogue scale The visual analogue scale is a measurement to assess the severity of pain. In this context, the patients will be assessed by letting them point the score on a device based on their pain experiences.
  The minimum value is 0 and the maximum is 10. The higher the score, the more severe the pain is.

SECONDARY OUTCOMES:
Pain within 2 hours after non obstetric lower abdominal surgerysurgery: visual analogue scale | 2 hours after surgery
  Measured by visual analogue scale The visual analogue scale is a measurement to assess the severity of pain. In this context, the patients will be assessed by letting them point the score on a device based on their pain experiences.
  The minimum value is 0 and the maximum is 10. The higher the score, the more severe the pain is.
Pain within 6 hours after non obstetric lower abdominal surgerysurgery: visual analogue scale | 6 hours after surgery
  Measured by visual analogue scale The visual analogue scale is a measurement to assess the severity of pain. In this context, the patients will be assessed by letting them point the score on a device based on their pain experiences.
  The minimum value is 0 and the maximum is 10. The higher the score, the more severe the pain is.
Pain within 12 hours after non obstetric lower abdominal surgerysurgery: visual analogue scale | 12 hours after surgery
  Measured by visual analogue scale The visual analogue scale is a measurement to assess the severity of pain. In this context, the patients will be assessed by letting them point the score on a device based on their pain experiences.
  The minimum value is 0 and the maximum is 10. The higher the score, the more severe the pain is.
Cumulative morphine requirement within 2 hours after non obstetric lower abdominal surgery | 2 hours after surgery
  Measured by total consumption of morphine on patient controlled analgesia machine
Cumulative morphine requirement within 6 hours after non obstetric lower abdominal surgery | 6 hours after surgery
  Measured by total consumption of morphine on patient controlled analgesia machine
Cumulative morphine requirement within 12 hours after non obstetric lower abdominal surgery | 12 hours after surgery
  Measured by total consumption of morphine on patient controlled analgesia machine

CONTACTS AND LOCATIONS:
Locations (1):
- Cipto Mangunkusumo Cental National Hospital, Jakarta, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Weiser TG, Regenbogen SE, Thompson KD, Haynes AB, Lipsitz SR, Berry WR, Gawande AA. An estimation of the global volume of surgery: a modelling strategy based on available data. Lancet. 2008 Jul 12;372(9633):139-144. doi: 10.1016/S0140-6736(08)60878-8. Epub 2008 Jun 24. PMID 18582931
- [Result] Bruce J, Quinlan J. Chronic Post Surgical Pain. Rev Pain. 2011 Sep;5(3):23-9. doi: 10.1177/204946371100500306. PMID 26526062
- [Result] Ip HY, Abrishami A, Peng PW, Wong J, Chung F. Predictors of postoperative pain and analgesic consumption: a qualitative systematic review. Anesthesiology. 2009 Sep;111(3):657-77. doi: 10.1097/ALN.0b013e3181aae87a. PMID 19672167
- [Result] Shavit Y, Fridel K, Beilin B. Postoperative pain management and proinflammatory cytokines: animal and human studies. J Neuroimmune Pharmacol. 2006 Dec;1(4):443-51. doi: 10.1007/s11481-006-9043-1. Epub 2006 Sep 29. PMID 18040817
- [Result] Beilin B, Shavit Y, Trabekin E, Mordashev B, Mayburd E, Zeidel A, Bessler H. The effects of postoperative pain management on immune response to surgery. Anesth Analg. 2003 Sep;97(3):822-827. doi: 10.1213/01.ANE.0000078586.82810.3B. PMID 12933409
- [Result] Lee BH, Park JO, Suk KS, Kim TH, Lee HM, Park MS, Lee SH, Park S, Lee JY, Ko SK, Moon SH. Pre-emptive and multi-modal perioperative pain management may improve quality of life in patients undergoing spinal surgery. Pain Physician. 2013 May-Jun;16(3):E217-26. PMID 23703420